CLINICAL TRIAL: NCT05945693
Title: Role of Specialized Pro-resolving Mediators on Inflammation, Cardiometabolic Health, Disease Progression, and Quality of Life in Patients With Rheumatoid Arthritis After Omega-3 PUFA Supplementation and Aerobic Exercise Training.
Brief Title: Omega-3 and Exercise in Rheumatoid Arthritis People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Ciencias de la Salud, Universidad de O'Higgins (Other)
Collaborators: Universidad Nacional Andres Bello (Other); University of Manitoba (Other); University of Guelph (Other); University of Chile (Other)
Responsible Party: Principal Investigator, Sebastian Jannas-Vela, Assistant Professor, Instituto de Ciencias de la Salud, Universidad de O'Higgins
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 11220333
Record Dates: First submitted 2023-07-03; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: omega-3; exercise; oxylipins; specialized pro-resolving mediators; inflammation; gene expression
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Inflammation | interventions — Docosahexaenoic Acids; Exercise

STUDY DESIGN:
Intervention Model Description: This study consists of a 16-week intervention with omega-3 polyunsaturated fatty acids (n-3 PUFAs) and/or aerobic exercise (AEx) training. The subjects will be randomly assigned in a double-blinded manner to one of four groups: placebo control (PLA), PLA+AEx, n-3, or n-3+AEx. The training sessions will be conducted at the Laboratorio de Ciencias del Ejercicio en el Ciclo Vital (Lab-CERVITAL), Universidad de O'Higgins. The week before intervention the participants will perform RA-specific tests (e.g., Disease Activity Score-28) and functional measurements (e.g., handgrip strength), peak aerobic capacity test, a dietary and physical activity assessment, and blood samples will be collected. Subsequently, participants will start their 16-week intervention (PLA, PLA+AEx, n-3, or n-3+AEx). At the end of the intervention the same initial measurements, questionnaires, and assessments will be collected.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking process will ensure that both the participants and the investigators involved in the study remain unaware of the treatment assignments throughout the entire duration of the study. A unique identification code will be assigned to each participant upon enrollment, which conceals their treatment allocation. The allocation sequence will be generated by a person not directly involved in the study. The capsules in the experimental intervention and the control treatment, will be packaged identically to maintain visual similarity. The packaging materials and labeling will be designed to be indistinguishable between the two groups. In addition, all outcome assessments and data collection procedures will be performed by personnel who are blinded to the treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo control (Placebo Comparator): The participants will be supplemented with 5 capsules per day of a placebo-filled gelatin capsule.
  Interventions: Dietary Supplement: Placebo
- Placebo and aerobic exercise (Active Comparator): The participants will be supplemented with 5 capsules per day of a placebo-filled gelatin capsule and will perform aerobic type exercise training three times per week, on non-consecutive days, with a total time of 20-60 minutes per day.
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Aerobic exercise
- Omega-3 (Experimental): The participants will be supplemented with 5 capsules per day of Omega UP (Newscience, Chile) equivalent to 2.5 g/d of DHA and 0.5 g/d of EPA.
  Interventions: Dietary Supplement: Omega-3
- Omega-3 and aerobic exercise (Experimental): The participants will be supplemented with 5 capsules per day of Omega UP (Newscience, Chile) equivalent to 2.5 g/d of DHA and 0.5 g/d of EPA and will perform aerobic type exercise training three times per week, on non-consecutive days, with a total time of 20-60 minutes per day.
  Interventions: Dietary Supplement: Omega-3; Dietary Supplement: Aerobic exercise

INTERVENTIONS:
Dietary Supplement: Placebo — The participants will be supplemented with 5 capsules per day of a placebo-filled gelatin capsule for 16 weeks.
  Arms: Placebo and aerobic exercise; Placebo control
Dietary Supplement: Omega-3 — The participants will be supplemented with 5 capsules per day of Omega UP (Newscience, Chile) equivalent to 2.5 g/d of DHA and 0.5 g/d of EPA for 16 weeks.
  Arms: Omega-3; Omega-3 and aerobic exercise
Dietary Supplement: Aerobic exercise — The participants will perform aerobic-type exercise training three times per week, on non-consecutive days, with a total time of 20-60 minutes per day for 16 weeks.
  Arms: Omega-3 and aerobic exercise; Placebo and aerobic exercise

SUMMARY:
Rheumatoid arthritis (RA) is a chronic inflammatory disease characterized by autoantibody production and synovial membrane damage. It significantly impairs overall function and quality of life. Consumption of omega-3 (n-3) polyunsaturated fatty acids (PUFAs) and regular aerobic exercise (AEx) training are reported to have positive effects on the progression of RA. However, the mechanisms behind these benefits are still inconclusive. This study aims to investigate the effects of n-3 PUFA supplementation and AEx training on disease progression, cardiometabolic health, and quality of life, and their association with the plasma and synovial fluid levels of specialized pro-resolving mediators (SPMs) in subjects with RA. The study consists of a 16-week intervention period, during which participants will be randomly assigned in a double-blinded manner to one of four groups: placebo control (PLA), PLA+AEx, n-3, or n-3+AEx. The PLA groups will be given a gelatin-filled capsule, while the n-3 groups will be given n-3 PUFAs equivalent to 2.5 g/d of docosahexaenoic acid and 0.5 g/d of eicosapentaenoic acid. The AEx groups will exercise thrice per week on a stationary electronically braked cycle ergometer at 60-70% of their VO2peak for 50-60 minutes. Before and after the intervention, participants will undergo RA-specific and functional measurements, peak aerobic capacity test, and a dietary and physical activity assessment. Venous blood and synovial fluid from the knee joint will be collected. Changes in disease progression, cardiometabolic health, quality of life, and erythrocyte membrane composition to assess n-3 incorporation, SPM levels, inflammatory markers, and gene expression from blood and synovial fluid will be analyzed. The study aims to elucidate the SPMs that regulate the inflammatory gene expression pathways and associate them with improvements in disease progression, cardiometabolic health, and quality of life after n-3 PUFA supplementation and AEx training.

DETAILED DESCRIPTION:
Research hypothesis: N-3 PUFA and AEx will have synergistic effects on disease progression, cardiometabolic health, and quality of life in individuals with RA, and these changes will be associated with SPM production in blood and synovial fluid.

General aim: To investigate the effects of n-3 PUFA supplementation and AEx training on disease progression, cardiometabolic health, and quality of life and their association with the plasma and synovial fluid levels of SPMs in individuals with RA.

Specific aims:

1. To compare the effects of n-3 PUFA supplementation, AEx training, and the combination of both on disease progression, cardiometabolic health, and quality of life in individuals with RA.
2. To compare the effects of n-3 PUFA supplementation, AEx, and the combination of both on the plasma and synovial fluid levels of the SPMs in individuals with RA.
3. To examine the relationship between the plasma levels of the n-3 PUFA derived SPMs with systemic disease progression, cardiometabolic health, and quality of life in individuals with RA

Study design 88 Participants will be recruited from hospitals and private clinics in the central region of Chile, whereas all the interventions regarding AEx will be carried out at the Universidad de O'Higgins and the Hospital Regional de Rancagua. All institutions are in the Región del Libertador Bernardo O'Higgins, Chile. This study consists of a 16-week intervention with n-3 PUFAs and/or aerobic exercise (AEx) training. The subjects will be randomly assigned in a double-blinded manner to one of four groups: placebo control (PLA), PLA+AEx, n-3, or n-3+AEx. A stratified randomized assignment (by block) process will be employed to ensure that the experimental groups are balanced for disease activity, pharmacological treatment, sex, and age. The training sessions will be conducted at the Laboratorio de Ciencias del Ejercicio en el Ciclo Vital (Lab-CERVITAL), Universidad de O'Higgins. The week before intervention the participants will perform RA specific tests (e.g., Disease Activity Score-28) and functional measurements (e.g., handgrip strength), peak aerobic capacity test, a dietary and physical activity assessment, and blood samples will be collected. Subsequently, participants will start their 16-week intervention (PLA, PLA+AEx, n-3, or n-3+AEx). At the end of the intervention the same initial measurements, questionnaires, and assessments will be collected. In a subgroup of participants (n=24 in total or n=6 per group) extraction of synovial fluid will be performed before and after the intervention.

The participants will be supplemented with either 5 capsules per day of Omega UP (Newscience, Chile) equivalent to 2.5 g/d of DHA and 0.5 g/d of EPA or a placebo filled gelatin capsule. The current doses are within the limits recommended by the European Food Safety Authority and have been shown to be safe, to be incorporated into cell membranes, and to produce significant improvements in overall health in individuals with RA. Capsules will be placed into de-identified bottles by people not involved in the study and provided to the participants to ensure double blinding. The exercise intervention will be performed according to the recommendations from the European Alliance of Associations for Rheumatology (EULAR) consisting of aerobic type exercise training three times per week, on non-consecutive days, with a total time of 20-60 minutes. The AEx will be performed on a stationary electronically braked cycle ergometer starting at 40-50% of VO2peak for 20 minutes. The intensity and volume of cycling will then be gradually increased to target at least 60-70% of VO2peak for 50-60 minutes over the final 10 weeks. Heart rate, power output and rating of perceived exertion (RPE) will be monitored during training intervention.

Statistical analysis Results will be expressed as mean ± SD. A two-way ANOVA with repeated measures followed by Fisher's least significant difference post-test for multiple comparisons between groups will be used. Linear regression models will be constructed to examine the association between SPMs and clinical, functional, and health parameters, accounting for participant age, sex, and BMI as covariates. A value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis with moderate disease activity as defined by the Disease Activity Score 28 (DAS28) > 2.6 and < 5.1.
* Participants taking nonsteroidal anti-inflammatory drugs (NSAIDs), glucocorticoids, or disease-modifying anti-rheumatic drugs (DMARDs) will be eligible; however, the dosages of these agents must be constant at least four weeks before, must remain within this limit throughout the study, and prednisone dose should not be higher than 7.5 mg/d

Exclusion Criteria:

* Individuals diagnosed with gastrointestinal or metabolic diseases, regular alcohol abuse, smokers, and dietary supplement intake (e.g., fish oil capsules) or consumption of fish > 2 times per week.
* Individuals that perform regular aerobic exercise (> 150 min moderate intensity per week) or have any physical or biomechanical limitations to complete the exercise program
* Individuals that present blood levels of aspartate aminotransferase, alanine transaminase, or creatinine higher than 1.5 times the maximum normal limit and total bilirubin levels of more than 1.8 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Early morning stiffness | Pre and post intervention (16 weeks)
  Duration of morning stiffness in minutes

SECONDARY OUTCOMES:
Disease activity score-28 | Pre and post intervention (16 weeks)
  Severity of rheumatoid arthritis using clinical and laboratory data
Health assessment questionnaire disability index | Pre and post intervention (16 weeks)
  Questionnaire that evaluates the functional status of individuals with rheumatoid arthritis
Quality of life RA | Pre and post intervention (16 weeks)
  8-item RA-specific health-related quality of life instrument scale.
Analgesic use | Pre and post intervention (16 weeks)
  Pill counts for paracetamol and NSAIDs
Timed Up and Go test | Pre and post intervention (16 weeks)
  The participant starts in a seated position, stands up upon command, walks 3 meters, turns around, walks back to the chair, and sits down. The time stops when the subject is seated
Short Physical Performance Battery | Pre and post intervention (16 weeks)
  Evaluates lower extremity functional performance using timed measures of standing balance, a 4-meter walk, and five repetitive chair stands
Handgrip strength | Pre and post intervention (16 weeks)
  Measures the maximum isometric strength of the hand and forearm muscles.
Peak aerobic capacity | Pre and post intervention (16 weeks)
  Incremental cycling test to exhaustion using a recumbent cycle ergometer to measure aerobic capacity.
Dietary assessment | Pre and post intervention (16 weeks)
  Dietary record using image-assisted method over three days (two consecutive weekdays and one weekend day)
Global Physical Activity Questionnaire | Pre and post intervention (16 weeks)
  Questionnaire to assess physical activity levels
Plasma rheumatoid factor | Pre and post intervention (16 weeks)
  Plasma rheumatoid factor will be measured via commercial ELISA assay kits.
Total cholesterol | Pre and post intervention (16 weeks)
  Total cholesterol will be measured.
LDL cholesterol | Pre and post intervention (16 weeks)
  LDL cholesterol will be measured.
HDL cholesterol | Pre and post intervention (16 weeks)
  HDL cholesterol will be measured.
TNF-alfa | Pre and post intervention (16 weeks)
  Plasma TNF-alfa will be measured via commercial ELISA assay kits.
IL-10 | Pre and post intervention (16 weeks)
  Plasma IL-10 will be measured via commercial ELISA assay kits.
Gene expression | Pre and post intervention (16 weeks)
  Real-time PCR will be carried out to quantify the changes in the expression of genes associated with inflammatory pathways and oxylipin synthesis
Phospholipid fatty acid composition | Pre and post intervention (16 weeks)
  Quantitative extraction of total lipids from erythrocytes, plasma, and synovial fluid will be carried out.
Oxylipin analyses | Pre and post intervention (16 weeks)
  Plasma and synovial fluid samples will be analyzed in duplicate for oxylipins by HPLC/MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Jannas-Vela, PhD, Principal Investigator — Universidad de O'Higgins
Locations (1):
- Universidad de O'Higgins, Rancagua, Libertador Bernardo O'Higgins, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jannas-Vela S, Candia AA, Penailillo L, Barrios-Troncoso P, Zapata-Urzua J, Rey-Puente J, Aukema HM, Mutch DM, Valenzuela R, Valladares-Ide D. Role of specialized pro-resolving mediators on inflammation, cardiometabolic health, disease progression, and quality of life after omega-3 PUFA supplementation and aerobic exercise training in individuals with rheumatoid arthritis: a randomized 16-week, placebo-controlled interventional trial. F1000Res. 2023 Aug 7;12:942. doi: 10.12688/f1000research.138392.1. eCollection 2023. PMID 38778807